CLINICAL TRIAL: NCT02234154
Title: A Study to Evaluate the Safety and Effectiveness of the TOPS System
Brief Title: Post-market Study of the TOPS™ System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Premia Spine (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1513-CL-TP-01 NOT UK
Record Dates: First submitted 2014-09-04; First posted 2014-09-09 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-04

CONDITIONS: Lumbar Spinal Stenosis; Spondylolisthesis
MeSH Terms: conditions — Spinal Stenosis; Spondylolisthesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TOPS System (Other): Post Marketing Study
  Interventions: Device: TOPS System

INTERVENTIONS:
Device: TOPS System — Non-randomized study involving implantation of a TOPS via lumbar surgery to decompress and provide stability to the index level.

SUMMARY:
This Single-Arm Post-Marketing Evaluation will gauge the improvement in function and pain for lumbar spinal stenosis and spondylolisthesis patients with the TOPS System.

DETAILED DESCRIPTION:
This study is being conducted to evaluate the TOPS™ SP System from ("TOPS™ System" or "TOPS"). TOPS is an alternative to spinal fusion and is designed to stabilize but not fuse the affected vertebral level to alleviate pain stemming from degenerative spondylolisthesis (abnormal/excessive movement of the vertebrae causing pain in the lower back and legs) and spinal stenosis (narrowing of the spinal canal resulting in compression of nerves producing symptoms of pain, numbness and tingling in the legs).

ELIGIBILITY:
IInclusion Criteria - Prospective subjects must meet all of the following criteria to be considered eligible for inclusion in this clinic study:

* Age 40-85 years old;
* One or both of the following at a single level from L3 to L5; (1) symptomatic monosegmental lumbar spinal stenosis or facet arthrosis, (2) degenerative spondylolisthesis up to and including grade 1.
* At least three (3) months of failed, conservative treatment prior to surgery (unless deemed inadvisable due to progressive motor weakness or other evidence of rapidly deteriorating condition) including the use of anti-inflammatory medications at maximum specified dosage, administration of epidural/facet injections, rest, heat, electrotherapy and/or physical therapy;
* Narrowing of the lumbar spinal canal (central and/or foramenal) classified as moderate to severe using CT scans/MRI;
* VAS leg pain of at least 40/100;
* Oswestry Disability Index score of at least 40/100;
* Lower back pain or sciatica with or without spinal claudication and
* Psychosocially, mentally and physically able to fully comply with the clinical protocol and willing to adhere to follow-up schedule and requirements.

Exclusion Criteria - Prospective subjects must not meet any of the exclusion criteria to participate in this clinical study:

* Primary diagnosis of discogenic back pain at the TOPS System level;
* Back or non-radicular leg pain of unknown etiology at the index level;
* Lytic spondylolisthesis at the index level;
* More than one (1) motion segment involved in the degenerative pathology to the extent that justifies its inclusion in the surgical procedure, unless a decompression alone can be done at that level without compromising stability;
* Known allergy to titanium and/or polyurethane;
* Supplemental interbody support required (e.g., bone graft, spacers, VBRs, or fusion cages) at the index level;
* Clinically compromised vertebral bodies at the affected level(s) due to any traumatic, neoplastic, metabolic or infectious pathology;
* Deformity of the spine that would compromise the implant, e.g. scoliosis of greater than ten (10) degrees;
* Morbid obesity defined as a body mass index > 40 or a weight more than 100 lbs. over ideal body weight;
* DEXA bone density measured T score equal to or lower than - 2.0;
* Paget's disease, osteomalacia, osteogenesis imperfecta, thyroid and/or parathyroid gland disorder and/or any other metabolic bone disease;
* Active infection;
* AIDS, HIV, or active hepatitis;
* Rheumatoid arthritis or other autoimmune disease;
* Tuberculosis active or in the past 3 years;
* Active malignancy: unless treated with curative intent and there have been no clinical signs or symptoms of the malignancy for at least 5 years;
* Medical condntions requiring treatment with any drugs known to potentially interfere with bone/soft tissue healing;
* Pregnant or interested in becoming pregnant in the next 3 years;
* Current chemical/alcohol dependency or significant psychosocial disturbance;
* Cauda equina syndrome or neurogenic bowel/bladder dysfunction;
* Severe arterial insufficiency of the legs, peripheral vascular disease;
* Sustained pathologic fractures of the vertebra or multiple fractures of the vertebra or hip;
* Significant peripheral neuropathy;
* Immunologically suppressed, received steroids > 1 month out of the past year;
* Insulin-dependent diabetes mellitus;
* Life expectancy less than 3 years;
* Waddell signs > 3;
* Currently involved in active spinal litigation OR
* Subject is incarcerated.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-12; Primary Completion 2017-03 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Improvement in ODI and Improvement in VAS leg score v | 24 months post implantation
  Composite endpoint - Subjects who exhibit a reduction of 15 percent in their Oswestry Disability Index (ODI) score compared to their preoperative ODI score AND a reduction of at least 20mm (20% improvement) in either of their VAS Leg Score will be considered a success.

SECONDARY OUTCOMES:
Improvement in back and leg visual analog scales (VAS) | 24 month postoperatively
  A failure to meet of any of the secondary endpoints will not be considered a therapeutic failure unless such a failure requires subsequent surgical intervention.
Improvement in ZCQ scores | 24 months postoperatively
  A failure to meet of any of the secondary endpoints will not be considered a therapeutic failure unless such a failure requires subsequent surgical intervention.
Quality of life (SF-36) | 24 months postoperatively
  A failure to meet of any of the secondary endpoints will not be considered a therapeutic failure unless such a failure requires subsequent surgical intervention.
Maintenance or improvement in neurological symptoms | 24 months postoperatively
  A failure to meet of any of the secondary endpoints will not be considered a therapeutic failure unless such a failure requires subsequent surgical intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Masood Shafafy, MD, Principal Investigator — Queens Medical Centre Nottingham
Locations (1):
- Queens Medical Centre, Nottingham, Nottinghamshire, United Kingdom